CLINICAL TRIAL: NCT05676125
Title: Trunk Muscle Strength and Endurance in Chronic Ankle Instability
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, noha mahmoud youssef aboelezz, Assistant Lecturer, Cairo University
Other Study IDs: P.T.REC/012/003263
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Chronic Ankle Instability
Keywords: CAI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic ankle instabilty group: females with previous history of ankle sprain
- control group: healthy feamles

SUMMARY:
Evaluation of trunk muscle strength in patients of chronic ankle instability

DETAILED DESCRIPTION:
This study will be conducted in the Isokinetic Laboratory. Sixty females with CAI will participate in this study. Their age will range from 18-30 years. They will be divided into two groups; the experimental and the control group. The experimental group will involve 30 females with CAI and the control group will involve 30 healthy females. The isokinetic strength of trunk muscles will be evaluated in a concentric mode of muscle contraction at an angular velocity 60°/sec. McGill test will be used to assess trunk muscle endurance.

ELIGIBILITY:
Inclusion Criteria:

* The initial sprain must have occurred at least 12 months prior to study enrollment.
* The most recent injury must have occurred more than three months prior to study enrollment (unassisted walking without limping for at least three months after injury).
* A history of the previously injured ankle joint giving way, recurrent sprain and/or feelings of instability.
* The injured/unstable ankle functionally weaker, more painful, looser, and less functional than the uninvolved ankle.
* The Oswesty Disability Index (ODI) score for both groups is from 0 to 20% (minimal disability) (Fairbank and Pynsent, 2000).

6- The Identification of Functional Ankle Instability questionnaire (IdFAI) score is less than 10 for the experimental group and 11 or more for the control group (Simon et al., 2012).

Exclusion Criteria:

* 1-A history of previous surgeries or fractures in either limb of lower extremity.

  2-Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous three months, which impacted joint integrity and function (ie, sprains, fractures) resulting in at least one interrupted day of desired physical activity.

  3-Any positive ﬁndings of the anterior drawer or talar tilt test (Hubbard and Kaminski, 2002).

  4-Any shoulder (Kibler et al., 2006) or elbow injuries (Ben Kibler and Sciascia, 2004).

Ages: 18 Years to 30 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — females are at higher risk than male
Study Population: faculty of physical therapy outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
trunk muscles strength | this will be evaluated on day one
  concentric peak torque of trunk flexors and extensors
core muscle endurance | this will be evaluated on day one
  mcgill core endurance tests

CONTACTS AND LOCATIONS:
Overall Officials: salam M Elhafez, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Dokki, Egypt